CLINICAL TRIAL: NCT02671448
Title: Pilot Trial of Homebound Stem Cell Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Screening
Other Study IDs: 15-022
Record Dates: First submitted 2016-01-28; First posted 2016-02-02 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Plasma Cell Dyscrasia
Keywords: Homebound; Homecare; 15-022
MeSH Terms: conditions — Paraproteinemias | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Intervention Model Description: This pilot trial will be the first attempt at developing a homebound hematopoietic stem cell transplant (HSCT) program at MSK.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Homebound After Stem Cell Transplantation (Experimental): The primary research outputs and measurements are the instruments/surveys, assessments, and video diaries to be completed by the patients, their caregivers and the healthcare providers during the time of the home transplantation care. Protocol-specific interventions during homebound care will continue until patient has achieved neutrophil engraftment. Post engraftment, standard of care practice will resume. Once discharged from homebound care, the patient will complete routine post-HSCT follow-up visits in the clinic setting.
  Interventions: Behavioral: Home monitoring teleconsult visits; Behavioral: Patient Reported Outcomes (PRO); Behavioral: Caregiver Reported Outcomes instruments

INTERVENTIONS:
Behavioral: Home monitoring teleconsult visits — A tablet will be provided to both the patient and the caregiver during the homecare portion of the study. The tablet will remain at the home, to be used by the patient and the caregiver during daily homecare visits to complete instruments/surveys and video diary recording sessions.
Behavioral: Patient Reported Outcomes (PRO) — Distress Thermometer, MSK-Modified M.D. Anderson Symptom Inventory (MDASI) Instrument, FACT-G Instrument, FACT-BMT Instrument
Behavioral: Caregiver Reported Outcomes instruments — Distress Thermometer, Caregiver Reaction Assessment (CRA) Instrument, The Caregiver Quality of Life Index-Cancer (CQOLC) Scale, Satisfaction Questionnaire, Video Diary Entries

SUMMARY:
In this study, the investigators plan to see what happens when a person receives care in the home setting. They want to find out if caring for a patient who has been treated with an ASCT in the home setting is feasible. They want to find out what effects good and/or bad this will have on the patient's recovery and treatment after ASCT. Studies in other institutions have shown that providing care in the home setting after ASCT is safe, increases patient satisfaction, and can decrease the risk of infection. It is our hope that this new approach of providing care in the home setting will prove to be a feasible and safe option for patients at Memorial Sloan Kettering Cancer Center (MSK).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Plasma cell dyscrasia
* Treatment plan including Autologous HSCT
* 18-80 years of age
* Appropriate homebound setting as defined by one of the following:

  * Lodging at the MSK Residence.
  * Staying at home or a "home equivalent" in any one of the zip codes as outlined in the appendix. Home equivalent is defined as a residence which may or may not be the primary residence of the patient.
  * "Home equivalent" must pass the "Home Environment Screening Tool" for homebound stem cell transplantation (not required for other MSK recognized lodging facility).
* Adequate caregiver support as defined by:

  * Single or multiple informal caregivers willing and able to provide 24 hour a day, seven day a week supervision of the transplant recipient in their home or "home-like" environment.
  * Caregiver willing and able to fulfill the basic stem cell transplant caregiver education requirements as determined by caregiver and healthcare team, including social worker
* Have Wi-Fi connection
* Appropriate third party payer coverage for "Homebound Stem Cell Transplant Program"
* Both patient and caregiver willing to give and sign informed consent.

Exclusion Criteria:

* Patients with a documented active infection prior to starting their preparative regimen. This includes grade 3 or higher viral, bacterial, or fungal infection.
* Uncontrolled arrhythmias
* Active or uncontrolled pulmonary disease
* Karnofsky Performance Scale (KPS) score <80
* Sorror Co-morbidity index ≥ 4 except in patients with history of resected cancers
* Creatinine clearance (calculated or measured) of < 50 cc/minute
* Inability of patient or caregiver to speak or read English (we currently do not have the manpower to translate nor staff a multilingual homebound stem cell transplant program with adequate educational materials).
* Inadequate housing arrangements
* Inadequate caregiver arrangements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2016-01; Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
readmission rate by 21 days post HSCT | 21 days post HSCT
  the homebound procedure will be considered promising if no more than 10 patients are readmitted to the hospital within 21 days.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Landau, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/